CLINICAL TRIAL: NCT03303703
Title: Partnering Physical and Emotional Fitness: Improving Cardiac Recovery With Training in Emotion Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Kelly Wierenga, Postdoctoral Fellow, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ANF6098
Record Dates: First submitted 2017-09-20; First posted 2017-10-06 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Disease; Myocardial Infarction
Keywords: cardiac rehabilitation
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual cardiac rehabilitation and social phone calls for attention control.
- Intervention (Experimental): RENEwS intervention is five 60-minute group educational sessions.
  Interventions: Other: RENEwS

INTERVENTIONS:
Other: RENEwS — The intervention participants will meet with a trained interventionist for five 60-minute sessions as a group (two groups of five participants each). In the sessions time will be divided between didactic presentation of material, active practicing of techniques, group work focused on case studies, and worksheets for further practice at home. Topics covered within the intervention include emotional awareness, balancing emotional and physical wellbeing, selecting and implementing emotion regulation strategies (such as situation selections, mindfulness, engagement/avoidance, reappraisal, and emotional sharing), and emotional monitoring.
  Arms: Intervention

SUMMARY:
Patients who have just experienced a first major cardiac event are at risk of experiencing heightened negative emotions, which further negatively impact self-management of health behaviors. For those patients in phase II cardiac rehabilitation, there is an opportunity to address physical and emotional wellbeing to optimize self-management of diet and exercise. This study will pilot test an intervention aimed at improving these patients' abilities to regulate their emotions as a mechanism to minimize psychological distress and improve self-management of diet and exercise, as well as improve quality of life. This innovative pilot will generate knowledge about the impact of emotion regulation in first event cardiac rehabilitation patients.

DETAILED DESCRIPTION:
Significance. For the over 900,000 Americans experiencing a first cardiac event annually, stress, depression, and anxiety complicate recovery. Emotional distress, such as depression, anxiety, and rumination, detracts from a patient's ability to self-manage health behaviors such as diet and exercise. Those patients engaged in cardiac rehabilitation (CR) programs are in a unique position to enhance their recovery, yet do not regularly receive training to regulate their emotions. Effective emotion regulation can diminish symptoms of emotional distress. Developing an effective repertoire of emotion regulation strategies may be an important mechanism to strengthen self-management behaviors and quality of life. By understanding the neuroscience behind the mechanism of emotion regulation, targeted intervention strategies may aid in improving self-management behaviors. The newly developed RENEwS (Regulating Emotions to improve self-management of Nutrition, Exercise, and Stress) intervention is specifically designed to improve emotion regulation in CR patients and targets strengthening the recently discovered neural network task differentiation (analytic and emotional processing). RENEwS focuses on teaching emotion regulation strategies relevant to older adults following a first cardiac health event.

Purpose. The goals of this pilot study are to assess the initial effects of the RENEwS program on 1) negative emotions, 2) self-management behaviors of diet and exercise, and 3) quality of life in CR patients following an acute cardiac event. A secondary goal of the proposed research is to explore the neurological (using fMRI) and psychological (emotion regulation) mechanisms through which the RENEwS intervention reduces negative emotions, increases healthy diet and exercise, and increases quality of life. Study aims are:

Aim 1: Determine feasibility, acceptability, and effect size of the RENEwS intervention.

Aim 2: Determine the effect of the RENEwS program on negative emotions (depressive symptoms, anxiety, and rumination), self-management behaviors (diet and exercise), and quality of life as compared to an attention control group.

Aim 3a: Examine the relationships between emotion regulation and 1) selected psychological factors (patient activation, self-efficacy, decision-making, and attention), 2) neural processing (brain activation/function and task switching), and 3) perceived stress.

Aim 3b: Examine the possible mediating effect of emotion regulation, psychological factors, neural processing, and stress on the effectiveness of the RENEwS intervention to reduce negative emotions, and to improve self-management behaviors and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CVD
* phase II CR initiated within the past 2 months
* planned 12 weeks of CR
* living independently
* at least 40 years of age

Exclusion Criteria:

* patients who do not speak English
* have experienced cardiac arrest
* have an implanted pacemaker or defibrillator
* not approved safe for exercise

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Quality of life will be assessed with the 29-item Perceived Health Status (PROMIS-29). This measure examines quality of life across chronic illness populations. Total score of the PROMIS-29 will be used in the analysis of quality of life.

SECONDARY OUTCOMES:
Change in Psychological symptoms- Depression | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Depression will be measured with the 16 item Quick Inventory of Depressive Symptomatology and PROMIS depression-4.
Change in Psychological symptoms- Anxiety | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Anxiety will be assessed using the 7 anxiety items from the short-form of the Depression Anxiety Stress Scale and the PROMIS anxiety-4.
Change in Psychological symptoms- Rumination | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Rumination will be measured with the 22-item Ruminative Responses Scale.
Change in Self-management behaviors- Diet | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Diet will be assessed with the Nutrient Data Systems Report is a 24-item recall delivered by a trained nutritionist. This recall provides detailed intake information about over 150 different nutrients as well as food groups.39 Analysis of aims will use total intake of sodium and lipids.
Change in Self-management behaviors- Exercise | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Exercise will be assessed with actigraphy. Intensity and number of minutes of exercise will be assessed over a three-day period using the Actigraph Active Living Protocol. Total number of minutes and number of minutes in moderate to high intensity of exercise will be used for analysis of study aims.
Change in Emotion regulation | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Emotion regulation will be measured with the 16-item Emotional Regulation Profile-Revised.
Change in Stress | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Stress will be measured with the 10-item Perceived Stress Scale(PSS). PSS items are on a 5-point Likert-type scale and include subjective statements related to stress experienced in the last 30 days.
Change in Patient Activation | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Patient activation will be measured with the 10-item Patient Activation Measure.
Change in Self-efficacy | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Self-efficacy will be measured with the 6-item Self Efficacy for Managing Chronic Disease scale.
Change in Neural Function Brain Activation | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Brain activation will be assessed using functional Magnetic Resonance Imaging (fMRI). Neural network differentiation will be assessed using passive viewing of video clips, each 23 seconds in length. Half of the video clips will assess analytic thinking, and half empathetic/emotional cognition. Brain activity associated with each of these conditions will be assessed relative to a resting baseline, achieved by including fixation conditions of the same length and frequency as the video stimuli. All stimuli are presented with EPrime psychology software.
Change in Decision making | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Decision making will be assessed with the Iowa gambling task. This task will be conducted to assess decision making with a real-life simulation. In this task participants select decks of cards with the goal of winning as much money as possible.
Change in Attention | baseline, after completion of standard of care cardiac rehabilitation, and 3 months after completion of standard of care cardiac rehabilitation (an average of 5 months).
  Attention will be measured with the 13 item Attention Function Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788